CLINICAL TRIAL: NCT01686373
Title: Transcranial Direct Current Stimulation and Aphasia Treatment Outcomes
Brief Title: Brain Stimulation and Aphasia Treatment
Acronym: tDCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Julius Fridriksson, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11560FA12; U01DC011739 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-18 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Aphasia
Keywords: Aphasia; Brain; Stimulation; Communication; Stoke; Post; Phase II Clinical Trial; Treatment; tDCS; Fridriksson
MeSH Terms: conditions — Aphasia; Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activa Dose II Real tDCS (Experimental): Actual delivery of electrical stimulation
  Interventions: Device: Activa Dose II Real tDCS
- Activa Dose II Sham tDCS (Placebo Comparator): Sham delivery of electrical stimulation
  Interventions: Device: Activa Dose II Sham tDCS

INTERVENTIONS:
Device: Activa Dose II Real tDCS — 20 minutes of 1 milliamp active tDCS per treatment day (15 total sessions)
  Arms: Activa Dose II Real tDCS
Device: Activa Dose II Sham tDCS — 20 minutes of sham stimulation per treatment day (15 total sessions)
  Arms: Activa Dose II Sham tDCS

SUMMARY:
The purpose of this study is to assess the changes in language processing of patients with chronic, post-stroke aphasia following the application of brain stimulation. The brain stimulation the investigators administer is called transcranial direct current stimulation (tDCS). It involves passing a weak electrical current through the brain between two electrodes in the form of damp sponges. One sponge will be placed over a specified area on the damaged left hemisphere, while the other sponge will be placed on the right scalp. Computer-controlled speech-language treatment will be administered during the application of tDCS.

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability in the United States. Approximately one-third of all strokes result in acute language impairment (aphasia), with approximately one-fifth suffering from chronic aphasia. Unfortunately, the prognosis for moderate to severe chronic aphasia remains grim, as current behavioral treatment approaches usually offer only limited-to-modest benefit. Recent advancements in understanding the relationship between low current electrical brain stimulation and cortical plasticity suggest that the effect of behavioral aphasia treatment could possibly be enhanced using anodal transcranial direct current stimulation (A-tDCS). Indeed, we have shown how A-tDCS can significantly boost the effect of behavioral aphasia treatment. Based on these results as well as our other studies aimed at understanding how favorable brain plasticity correlates with positive treatment outcome in aphasia, we propose to conduct a Phase II clinical trial utilizing a futility design. Consistent with the goals of Program Announcement PAR-08-204 by the National Institute on Deafness and Other Communication Disorders (NIDCD), we plan to "evaluate whether there is sufficient evidence of short term improvement in humans to justify a phase III trial."

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing and able to give informed consent.
2. Patients must be willing and able to comply with study requirements.
3. Patients must be between 25- and 80-years of age.
4. Patients must be native English speakers.
5. Patients must be pre-morbidly right-handed.
6. Patients must have sustained a one-time ischemic stroke in the left-hemisphere.
7. Patients must be greater than 6-months post-stroke.
8. Patients must have an aphasia diagnosis as confirmed by the Western Aphasia Battery-Revised.
9. Patients must be MRI-compatible (e.g., no metal implants, not claustrophobic, etc.).
10. Patients must achieve at least 65% accuracy on naming task during screening -

Exclusion Criteria:

1. History of brain surgery
2. Seizures during the previous 12 months
3. Sensitive scalp (per patient report)
4. Able to overtly name more than an average of 140 out of 175 items during the pre-treatment picture naming test (Philadelphia Naming Test) during Visits 2 or 3.
5. Unable to overtly name at least an average of 5 out of 80 items during the pre-treatment functional magnetic resonance imaging (fMRI) sessions during Visits 2 or 3.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Fridriksson, PhD, Principal Investigator — Director
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina (USC), Columbia, South Carolina

REFERENCES:
- [Derived] Fridriksson J, Rorden C, Elm J, Sen S, George MS, Bonilha L. Transcranial Direct Current Stimulation vs Sham Stimulation to Treat Aphasia After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2018 Dec 1;75(12):1470-1476. doi: 10.1001/jamaneurol.2018.2287. PMID 30128538
- See also: University of South Carolina Aphasia Laboratory — http://sph.sc.edu/comd/fridriks/

RESULTS

PARTICIPANT FLOW:
Groups:
- Activa Dose II Real tDCS: Actual delivery of electrical stimulation
  Activa Dose II Real tDCS
- Activa Dose II Sham tDCS: Sham delivery of electrical stimulation
  Activa Dose II Sham tDCS
Period: Overall Study
Arm/Group | Activa Dose II Real tDCS | Activa Dose II Sham tDCS
Started | 34 | 40
Received 15 Treatment Sessions | 33 | 39
Completed | 31 | 38
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Activa Dose II Real tDCS | Activa Dose II Sham tDCS | Total
Number analyzed (Participants) | 34 | 40 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 60 (10) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 24 | 28 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 27 | 35 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 40 | 74

OUTCOME MEASURES:

1. Primary Outcome: The Philadelphia Naming Test (PNT) Plus the Naming 80 (a Portion of the Trained Items).
Description: The PNT includes 175 items and has a minimum score of 0 (zero items named correctly) and a maximum score of 175 (all items named correctly). The Naming 80 includes a portion of the trained treatment items (N=80) with a minimum score of 0 (zero items named correctly) and a maximum score of 80 (all items named correctly). For both scales, higher values represent better outcome. The average of two administrations of the PNT were added to the the average of two administrations of the Naming 80 for both time points. The outcome measure is the change in that value (averaged PNT + averaged Naming 80) from baseline to immediately post-treatment. Only two timepoints are used for this calculation: baseline and immediately post-treatment.
Time Frame: Immediately post-treatment
Measure: Mean (95% Confidence Interval); unit: PNT and Naming 80 score
Arm/Group | Activa Dose II Real tDCS | Activa Dose II Sham tDCS
Number analyzed (Participants) | 34 | 40
PNT and Naming 80 score | 13.9 [9.0 to 18.7] | 8.2 [3.8 to 12.6]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected until immediate post treatment testing sessions (2 weeks), and serious adverse events were collected until end of study (24 weeks).
Arm/Group | Activa Dose II Real tDCS | Activa Dose II Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/40
Other Adverse Events (participants affected / at risk) | 3/34 | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activa Dose II Real tDCS (N=34) | Activa Dose II Sham tDCS (N=40)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activa Dose II Real tDCS (N=34) | Activa Dose II Sham tDCS (N=40)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2012-08-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT01686373/SAP_000.pdf
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT01686373/Prot_001.pdf